CLINICAL TRIAL: NCT06661876
Title: Cardiac RadiothErapy For hEart faiLure
Acronym: CREFEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S69569
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Non-ischemic Cardiomyopathy; Ischemic Cardiomyopathy
Keywords: external beam radiotherapy; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5Gy whole heart radiotherapy (Experimental)
  Interventions: Radiation: 5 Gray Whole Heart external beam radiotherapy

INTERVENTIONS:
Radiation: 5 Gray Whole Heart external beam radiotherapy — EBRT will be delivered with photon energies restricted to 6 Megavoltage (MV) using intensity modulated radiotherapy (IMRT) or Volumetric modulated arc therapy (VMAT). Patients will be treated with a single fraction treatment up to a dose of 5Gy prescribed to the 95% PTV-encompassing isodose line (PTVD95% ≥5Gy). The near-maximum dose is limited to 5.35Gy (PTV D2% ≤ 5.35Gy). The treatment can be performed both as an inpatient or outpatient procedure.

SUMMARY:
Preliminary data suggests that patients suffering from advanced refractory heart failure (HF) could benefit from single low dose whole heart external beam radiotherapy (EBRT).

Objective: To explore in our center the efficacy of administering a EBRT treatment of 5Gy to the whole heart in patients with advanced and refractory HF. The hypothesis is that 5Gy EBRT to the whole heart can improve the left ventricular ejection fraction (LVEF) of these patients by a clinically relevant 5%.

Main study endpoints: The primary aim is to explore the efficacy of EBRT treatment for advanced refractory HF. Secondary endpoints include an assessment of safety, overall survival, hospital admissions, late toxicity, quality of life and the effect of the treatment on other heart function indicators (left ventricular volumes, NT-proBNP, Troponine, High sensitive CRP).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Advanced refractory HF NYHA class II, III or IV
* Stable HF for the last 6 months with maximal guideline-directed HF therapy
* Ischemic or dilated cardiomyopathy
* LVEF at baseline ≤ 35%
* Ability to give a written informed consent and willingness to return for follow-up

Exclusion Criteria:

* Eligible or in consideration for heart transplantation
* Pregnancy or breastfeeding
* Previous radiotherapy with cardiac involvement
* Any condition that is deemed a contraindication in the judgment of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | Baseline, week 6, week 12, and 6 months
  The hypothesis, based on recent preclinical and clinical data, is that 5Gy whole heart radiotherapy in advanced refractory HF patients can improve the LVEF and increase QOL with a low to very low toxicity profile. The efficacy will be defined as an improvement of at least 5% of the LVEF over a period of 6 months.

SECONDARY OUTCOMES:
Acute toxicity | toxicity occurring within 30 days after the radiation treatment.
  The tolerable acute toxicity will be assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) (U.S. Department of Health and Human Services 2017). It is defined as toxicity occurring within 30 days after the radiation treatment.
All-cause mortality | 6 months after the radiation treatment
  Death from any cause within 6 months after treatment. The Kaplan-Meier method will be used to estimate overall survival (OS).
Heart failure hospitalisation | Within 6 months after the radiation treatment
  The number and length of hospitalization related to HF after treatment and within 6 months after treatment. HF-related admissions are defined as a hospital admission lasting for more than 24 h, with signs or symptoms of congestion necessitating an increase of the dose of loop diuretics.
Late toxicity | 30 days to 6 months after the radiation treatment
  Late toxicity is defined as toxicity occurring after at least 30 days to 6 months after the radiation treatment and will be assessed by the CTCAE v5.0.
Quality of life - SF-36 | Baseline, 6 weeks, 12 weeks, and 6 months
  Health related quality-of-life (QOL) will be measured based on the SF-36. The 36-Item Short Form Survey (SF-36) is a set of generic, coherent, and easily administered quality of life measures that rely on patient self-reporting. The SF-36 evaluates 8 domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scale values for each domain range from 0 to 100 where the higher score defines a more favorable health state.
Quality of life - MLWHF | Baseline, 6 weeks, 12 weeks, and 6 months
  Health related quality-of-life (QOL) will be measured based on the Minnesota Living with Heart Failure (MLWHF) questionnaire. The MLWHFis a valid and reliable instrument consisting of 21 items for measuring QOL in patients with HF. It covers various domains including physical, emotional, social, and mental aspects of living with heart failure. Each item is scored on a scale (usually 0 to 5 or 0 to 6), with higher scores indicating a greater impact.
NT-proBNP levels | Baseline, week 6, week 12, and 6 months
  N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) will be measured as a biomarker of cardiac stress and heart failure severity. Levels are determined using standardized immunoassays and reported in picograms per milliliter (pg/mL). Higher NT-proBNP values generally indicate worse cardiac function and are associated with increased risk of adverse outcomes, whereas lower values suggest improved cardiac status.
High-sensitive troponin levels | Baseline, 6 weeks, 12 weeks, and 6 months
  High-sensitivity cardiac troponin will be measured as a biomarker of myocardial injury. High-sensitivity troponin allow detection of very low concentrations and provide accurate quantification across a wide range. Elevated hs-cTn values are associated with acute or chronic myocardial injury and adverse cardiovascular outcomes, whereas stable or low levels indicate absence of significant myocardial damage.
High-sensitivity C-reactive protein | Baseline, 6 weeks, 12 weeks, and 6 months
  High-sensitivity C-reactive protein (CRP) will be measured as a biomarker of systemic inflammation. High-sensitivity assays enable accurate detection of low CRP concentrations, reported in milligrams per liter (mg/L), which can reflect low-grade inflammation. Elevated hs-CRP levels are associated with increased cardiovascular risk and adverse outcomes, while lower levels indicate a more favorable inflammatory profile.
Left ventricular volumes | Baseline, 6 weeks, 12 weeks, and 6 months
  Left Ventricular End-Diastolic Volume (LVEDV) and End-Systolic Volume (LVESV) will be measured by transthoracic echocardiography using the Simpson's biplane method. These indices provide quantitative measures of left ventricular size and systolic function. Increased LVEDV and LVESV may reflect adverse remodeling and impaired function, whereas lower or normalized values indicate improved ventricular performance.
Ventricular arrhythmia burden | Baseline, 6 weeks, 12 weeks, and 6 months
  Ventricular arrhythmia burden will be measured by the cardiac implantable electronic device by assessing the Premature Ventricular Complexes (PVCs) burden; non-sustained Ventricular Tachycardia (nsVT), defined as ≥3 consecutive ventricular beats lasting <30 seconds; and sustainedventricular arrhythmia, defined as ≥30 seconds or requiring device intervention. Arrhythmia burden will be reported as the number of episodes detected during the specified follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in the article (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after publication of the main results, for at least 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to the corresponding author. Access will be granted upon approval of a data use agreement.